CLINICAL TRIAL: NCT01697202
Title: Fatigue in Rheumatoid Arthritis - Longitudinal Study
Status: Completed | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: GoteborgU
Record Dates: First submitted 2012-08-29; First posted 2012-10-02 (Estimated); Last update posted 2014-02-20 (Estimated); Status verified 2014-02

CONDITIONS: Fatigue; Rheumatoid Arthritis
MeSH Terms: conditions — Fatigue; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- no intervention

SUMMARY:
To investigate how the fatigue vary over time in persons with rheumatoid arthritis (RA) and which factors that may influence the fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnose of RA, age 20-65 years,

Exclusion Criteria:

* other serious physical or mental illness

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with RA at the Rheumatology clinic at Sahlgrenska University hospital Gothenburg, Sweden
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Fatigue | 4 times during the course of the study up to one year
  patient administered questionnaire

SECONDARY OUTCOMES:
Pain | 4 times during the course of the study up to one year
  patient administered questionnaire
Activity limitations | 4 times during the course of the study up to one year
  patient administered questionnaire
Disease activity | 4 times during the course of the study up to one year
  Tender and swollen joint count, patient-rated global health, inflammation parameters (DAS-28)
Health related quality of life | 4 times during the course of the study upto one year
  patient administered questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden